CLINICAL TRIAL: NCT03968601
Title: Prediction of Post-operative Left Ventricular Dysfunction in Primitive, Chronic Mitral Regurgitation Surgery With Preserved Ejection Fraction, by Pre-operative Global Longitudinal Strain Measure
Brief Title: Use of Pre-operative Global Longitudinal Strain to Predict Post-operative Left Ventricular Dysfunction in Mitral Regurgitation Surgery
Acronym: DysPO IM
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2018 CLERFOND; 2018-A02476-49 (Other: 2018-A02476-49)
Record Dates: First submitted 2019-04-05; First posted 2019-05-30 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Severe Mitral Regurgitation; Preserved Ventricular Ejection Fraction
Keywords: Severe mitral regurgitation; Preserved ventricular ejection fraction; Global Longitudinal Strain; Post-operative ventricular dysfunction; Echocardiography; Mitral surgery
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Wound Healing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohorte 1: Severe primary chronic mitral regurgitation with preserved left ventricular ejection fraction.
  Interventions: Other: Mitral regurgitation surgery such as mitral valve replacement or repair

INTERVENTIONS:
Other: Mitral regurgitation surgery such as mitral valve replacement or repair — Mitral regurgitation surgery such as mitral valve replacement or repair. All kind of mitral regurgitation surgery: replacement or repair, by median sternotomy of minimally invasive surgery, with or without tricuspid plasty

SUMMARY:
Primary mitral regurgitation (MR) is the second most frequent valve disease requiring surgery and it is important to identify patients whose outcome could be improved with surgery by considering the risks and benefits.

The current guidelines recommend surgery in patients with symptomatic severe mitral regurgitation or in asymptomatic patients who develop early signs of left ventricular (LV) dysfunction as a result of the MR.

However, it remains difficult to determine optimal timing for surgery with the current guidelines.

Early-stage LV dysfunction with normal LVEF predicts post-operative LV decompensation and poor prognosis and longitudinal myocardial function is suitable for detection of minor myocardial damage in patients with MR.

Thus, inestigators want to study the value of LV global longitudinal strain (GLS) to predict postoperative LV dysfunction in patients with chronic severe MR and preserved pre-operative LVEF.

The principal aim is to prove that the optimal timing for surgery, in asymptomatic chronic severe primary MR with preserved LVEF, is before GLS alteration, and that investigators should not wait for LV dilatation of dysfunction.

DETAILED DESCRIPTION:
Primary mitral regurgitation (MR) is the second most frequent valve disease requiring surgery.

In these patients, mitral repair is associated with excellent outcomes in terms of post-operative left ventricular (LV) function, and long-term survival when performed before the onset of severe symptoms, LV dysfunction or dilatation, pulmonary hypertension, and atrial fibrillation.

Thus, it is important to identify patients whose outcome could be improved with surgery by considering the risks and benefits.

The current guidelines recommend surgery in patients with symptomatic severe mitral regurgitation or in asymptomatic patients who develop early signs of left ventricular (LV) dysfunction as a result of the MR. LV dysfunction has been defined as LV ejection fraction (EF) 30% to 60% and/or LV end-systolic dimension (ESD) up to 45 mm.

However, it remains difficult to determine optimal timing for surgery with the current guidelines.

LVEF and LVESD, parameters proposed in the guideline, are difficult to interpret due to the influence of hemodynamic parameters of MR.

In asymptomatic patients who consider undergoing surgery, LVESD is rarely more than 45 mm.

In addition, LVEF in patients with severe MR often remains normal or higher, and subclinical LV dysfunction might be masked due to MR lowering of LV afterload.

Early-stage LV dysfunction with normal LVEF predicts post-operative LV decompensation and poor prognosis.

Therefore, it is a great challenge to identify potential LV dysfunction at an early stage and to perform surgery to prevent the development of irreversible LV dysfunction in patients with chronic severe MR.

Longitudinal myocardial function has been considered more sensitive than radial function and is therefore suitable for detection of minor myocardial damage in patients with MR.

A 2017 study proved that pre-operative GLS ≤ -18.4% can predict a preserved post-operative LVEF >50%.

Therefore, invetsigators want to study the value of LV global longitudinal strain (GLS) to predict postoperative LV dysfunction in patients with chronic severe MR and preserved pre-operative LVEF.

The principal aim is to prove that the optimal timing for surgery, in asymptomatic chronic severe primary MR with preserved LVEF, is before GLS alteration, and that investigators should not wait for LV dilatation of dysfunction.

Thus, investigators will recruit patients before surgery, measuring GLS during pre-operative conventional echography, and follow-up patients at 8 days, 1 month and 6 months to determine whether LVEF is preserved or not.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 or 4, primary and chronic mitral regurgitation, going for a planned surgery, with pre-operative left ventricular ejection fraction > 60% and left ventricular end-systolic dimension < 45mm.
* Able to consent.
* With a National Social Security number.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with another form of cardiopathy, such as dilated or hypertrophic cardiomyopathy, ischemic or rhythmic cardiopathy.
  * Patients with another valvular heart disease, such as significant aortic regurgitation or stenosis and significant mitral stenosis.
  * Poor echogenicity, insufficient for the different measures.
  * Severe pulmonary disease, inducing pulmonary hypertension.
  * Other causes of pulmonary hypertension.
  * Patients included in other studies with interventions able to interfere with our measures.
  * Pregnant women.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Pre-operative global longitudinal strain rate among patients going for mitral surgery. | During pre-operative visit
  Pre-operative global longitudinal strain in patients going for mitral regurgitation surgery with preserved LVEF, measured by echocardiography.

SECONDARY OUTCOMES:
Functional impact in terms of walking distance. | This test will be realized during pre-operative visit and repeated at 1-month and 6-months visits.
  6 Minute Walk Distance
Measure Quality of life: Minnesota Living with Heart Failure Questionnaire (MLHFQ) | This test will be realized during pre-operative visit and repeated at 1-month and 6-months visits.
  Minnesota Living with Heart Failure Questionnaire (MLHFQ), evaluating : legs swelling, walking and working capacity, presence of sleeping or breathing disorders, difficulties for sport, hobbies or relationships, side effects from medications, psychologic and economic impact of the disease. The total score goes from 0 (best quality of life) to 105 (worse impact).
Dyspnoea | This test will be realized during pre-operative visit and repeated at 8-days, 1-month and 6-months visits.
  Use of the New York Heart Association (NYHA) Functional Classification.
Left ventricular function | This test will be realized during pre-operative visit and repeated at 8-days, 1-month and 6-months visits.
  Left ventricular ejection fraction by Simpson method.
All-cause mortality, as the total number of death during the follow-up | At 8 days, 1-month and 6-months
  all death reported
Cardiovascular mortality, as the number of death from cardiovascular disease during the follow up | At 8 days, 1-month and 6-months
  Death by myocardial ischemia or infarction, heart failure, cardiac arrest, or cerebrovascular accident.
Number of patients hospitalized due to heart failure during the follow up | At 8 days, 1-month and 6-months
  all re-hospitalisation reported
Pre-operative right ventricular function (measured by Tricuspid Annular Plane Systolic Excursion - TAPSE, Peak Systolic Velocity in DTI mode and Fractional Area Change). | These measures will be realized during pre-operative visit and repeated at 1-month and 6-months visits
  We aim to determine whether or not right ventricular function (measured by Tricuspid Annular Plane Systolic Excursion - TAPSE, Peak Systolic Velocity in DTI mode and Fractional Area Change) can have an impact on post-operative LVEF in patients going for mitral regurgitation surgery.
Pre-operative pulmonary arterial pressure determined by tricuspid regurgitation peak velocity | These measures will be realized during pre-operative visit and repeated at 1-month and 6-months visits.
  Ithe aim is to determine whether or not pulmonary hypertension (determined by tricuspid regurgitation peak velocity) can have an impact on post-operative LVEF in patients going for mitral regurgitation surgery.
Left ventricular ejection index | During pre-operative visit.
  Impact of this novel left ventricular ejection index (defined as indexed left ventricular end-systolic diameter divided by left ventricular outflow tract time-velocity integral) on post-operative left ventricular dysfunction, compared with global longitudinal strain.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Clerfond, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France